CLINICAL TRIAL: NCT01363544
Title: Train Your Brain? Exercise and Neurofeedback Intervention for ADHD
Brief Title: Train Your Brain and Exercise Your Heart? Advancing the Treatment for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: R. van Mourik (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Yulius (Unknown)
Responsible Party: Sponsor-Investigator, R. van Mourik, Dr, VU University of Amsterdam
Organization: VU University of Amsterdam (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZonMw 157003012
Record Dates: First submitted 2011-05-20; First posted 2011-06-01 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; neurofeedback; exercise; neurophysiology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity | interventions — Neurofeedback; Biofeedback, Psychology; Exercise; Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neurofeedback (Experimental)
  Interventions: Other: Neurofeedback
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- methylphenidate (Active Comparator): optimum dose of methylphenidate (assessed by a double blind placebo-controlled procedure)
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Other: Neurofeedback — 30 sessions of theta/beta neurofeedback within 10 weeks.
  Other Names: biofeedback
  Arms: Neurofeedback
Behavioral: Exercise — 30 sessions of individual sports training during 10 weeks.
  Other Names: sports
  Arms: Exercise
Drug: methylphenidate — The medication treatment is based on the MTA study and includes methylphenidate dosages of 5, 10, 15 (only for children with a weight below 25 kg) and 20 mg (only for children with a weight above 25 kg. The optimum dose will be determined by a double-blind placebo-controlled trial.
  Other Names: Not applicable, a generic form will be used.
  Arms: methylphenidate

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a developmental disorder that has a severe impact on a child's life and society. The core symptoms are attention problems, hyperactivity and impulsivity. These symptoms are related to disruptions in neurocognitive functions (such as inhibition: the ability to stop behavior) and disruptions in cortical regulation (such as 'cortical underarousal' as measured with the electroencephalogram). To date, the only evidence-based treatment is pharmacological. Medication is not effective in 20-30% of the children with ADHD and it can have side effects. The lack of alternatives for medication is a severe problem for these children and society.

Neurofeedback is becoming increasingly popular for treating ADHD. Neurofeedback is a training in which a person learns to alter its cortical regulation. Neurofeedback has been classified as 'probably effective' but its treatment effects need further empirical evidence. Non specific training effects, such as individual attention, may also contribute to treatment success. In this research project the investigators compare the efficacy of neurofeedback with exercise, a second non-pharmacological treatment, that may be comparable with neurofeedback in terms of non-specific effects. Exercise is also a promising treatment because of its positive effects on behavior, neurocognition in several patient groups. For these reasons, exercise deserves systematic research in ADHD. Furthermore, the investigators compare the efficacy of these two treatments with an optimal pharmacological treatment with methylphenidate (MPH). The main question is if neurofeedback and exercise are comparable in efficacy with MPH for treating ADHD. The primary outcome measure is behaviour (symptoms of ADHD). Secondary outcome measures include neurocognition and cortical regulation. This research project will give answer to the question if neurofeedback and exercise are as effective as MPH. Furthermore, it will give insight in how these interventions will give rise to improvements in behavior.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* IQ above 80

Exclusion Criteria:

* neurological disorder
* severe physical or cognitive disability

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2010-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Behaviour | Within 2 weeks after the end of treatment (T1) and 6 months after the end of treatment (T2)
  Behaviour is assessed with rating scales (SWAN, SDQ, SDSC,DCD) and actigraphy

SECONDARY OUTCOMES:
Improvement in neurocognition | Within 2 weeks after the end of treatment (T1) and 6 months after the end of treatment (T2)
  Neuorcognition is assessed with several neuropsychological tests measuring inhibition, working memory, time estimation and probabilistic learning
Improvement in neurophysiology | Within 2 weeks after the end of treatment (T1) and 6 months after the end of treatment (T2)
  Neurophysiology is measured with ERPs and quantitative EEG

CONTACTS AND LOCATIONS:
Overall Officials: Rosa van Mourik, PhD, Principal Investigator — VU University, faculty of psychology and education, department of clinical neuropsychology; Jaap Oosterlaan, Professor, Study Director — VU University, Faculty of Psychology and Education, department of clinical neuropsychology
Locations (6):
- Netherlands (6):
  - GGZ InGeest, Amsterdam, North Holland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Yulius voor Geestelijke Gezondheid, Rotterdam, South Holland
  - Stichting alles Kits, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Lucertis, Rotterdam, South Holland

REFERENCES:
- [Derived] Janssen TWP, Gelade K, Bink M, van Mourik R, Twisk JWR, Maras A, Oosterlaan J. Long-term effects of theta/beta neurofeedback on EEG power spectra in children with attention deficit hyperactivity disorder. Clin Neurophysiol. 2020 Jun;131(6):1332-1341. doi: 10.1016/j.clinph.2020.02.020. Epub 2020 Mar 12. PMID 32304847
- [Derived] Gelade K, Janssen TWP, Bink M, Twisk JWR, van Mourik R, Maras A, Oosterlaan J. A 6-month follow-up of an RCT on behavioral and neurocognitive effects of neurofeedback in children with ADHD. Eur Child Adolesc Psychiatry. 2018 May;27(5):581-593. doi: 10.1007/s00787-017-1072-1. Epub 2017 Nov 2. PMID 29098467
- [Derived] Janssen TWP, Bink M, Weeda WD, Gelade K, van Mourik R, Maras A, Oosterlaan J. Learning curves of theta/beta neurofeedback in children with ADHD. Eur Child Adolesc Psychiatry. 2017 May;26(5):573-582. doi: 10.1007/s00787-016-0920-8. Epub 2016 Nov 19. PMID 27866283
- [Derived] Gelade K, Janssen TW, Bink M, van Mourik R, Maras A, Oosterlaan J. Behavioral Effects of Neurofeedback Compared to Stimulants and Physical Activity in Attention-Deficit/Hyperactivity Disorder: A Randomized Controlled Trial. J Clin Psychiatry. 2016 Oct;77(10):e1270-e1277. doi: 10.4088/JCP.15m10149. PMID 27631143
- [Derived] Janssen TW, Bink M, Gelade K, van Mourik R, Maras A, Oosterlaan J. A Randomized Controlled Trial Investigating the Effects of Neurofeedback, Methylphenidate, and Physical Activity on Event-Related Potentials in Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2016 May;26(4):344-53. doi: 10.1089/cap.2015.0144. Epub 2016 Jan 15. PMID 26771913
- [Derived] Janssen TW, Bink M, Gelade K, van Mourik R, Maras A, Oosterlaan J. A randomized controlled trial into the effects of neurofeedback, methylphenidate, and physical activity on EEG power spectra in children with ADHD. J Child Psychol Psychiatry. 2016 May;57(5):633-44. doi: 10.1111/jcpp.12517. Epub 2016 Jan 8. PMID 26748531
- See also: sponsor website — http://www.zonmw.nl/
- See also: organization/sponsor website — http://www.yulius.nl